CLINICAL TRIAL: NCT02088671
Title: A Prospective, Blinded, Clinical Study for Assessing the Effectiveness of the NeuroSENSE for Monitoring the Hypnotic Depth of Anesthesia (DOA)
Brief Title: Effectiveness of the NeuroSENSE for Monitoring the Hypnotic Depth of Anesthesia
Status: Completed | Type: Observational
Sponsor: NeuroWave Systems Inc. (Industry)
Collaborators: U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency); Fraser Health (Other)
Responsible Party: Sponsor
Other Study IDs: 925-0701-DCI; W81XWH-06-C-0016 (Other Grant/Funding Number: US Army Medical Research Acquisition Activity)
Record Dates: First submitted 2014-03-12; First posted 2014-03-17 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Depth of Anesthesia (DOA)
Keywords: NeuroSENSE; Anesthesia; Hypnosis; Desflurane; Propofol
MeSH Terms: interventions — Desflurane; Propofol; Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Anesthesia: A single study group undergoing general anesthesia procedure to observe post-hoc the effect on the NeuroSENSE monitor readings.
  Interventions of interest:
  Drug: Propofol induction followed by randomized doses of desflurane; Emergence by stepping down the desflurane ET - See intervention descriptions.
  Device: Recording of EEG using NeuroSENSE (blinded to clinicians) - See intervention descriptions.
  Other: Data Collection - See intervention descriptions
  Interventions: Drug: Propofol induction followed by randomized doses of desflurane; Device: Recording of EEG using NeuroSENSE; Other: Data collection; Other: Drug: Emergence by stepping down the desflurane ET

INTERVENTIONS:
Drug: Propofol induction followed by randomized doses of desflurane — Anesthesia in all patients will be induced with iv propofol 1.5 mg/kg with extra 0.5 mg/kg doses as needed. Anesthesia will be maintained using inhaled desflurane in oxygen/air with the initial desflurane concentration of 1.2 MAC, which will be changed in steps of ±0.4 MAC after reaching the post-intubation steady state. The step changes will be initiated every 7.5 min, as follows: at every level of MAC there is a 1/3 chance in remaining at this level and a 2/3 chance of changing it. The anesthesiologist can accept the change to move to the new level. However, he/she can also reject it to remain at the current level for another 7.5 min. This scheme yields 3 possible desflurane levels: 0.8, 1.2 and 1.6 MAC. The anesthesiologist can also leave the randomization schedule at anytime if clinically indicated, and later re-start it at his/her discretion. All anesthetic doses and their changes fall within conventional dosing.
  Other Names: Suprane; Diprivan
Device: Recording of EEG using NeuroSENSE — The NeuroSENSE NS-701 system is a 2-channel device for brain activity monitoring in the operating room, intensive care unit, emergency room and other clinical settings. The system acquires and processes electroencephalograms (EEGs) via noninvasive electrodes placed on a patient's forehead. The acquired raw EEG signals and processed EEG variables are continuously displayed for interpretation by the clinician.
  The proprietary processed variable, WAVcns, quantifies the patient's brain activity, which is typically affected by anesthetic drugs. The system displays processed variables based on 2 bilateral channels (1 per brain hemisphere) for use as a supplement to the anesthesia standard of care.
  Note: the indications provided by the NeuroSENSE monitor are not used for anesthesia dosing or patient assessment in this study, and the anesthesia provider is blinded to the monitor readings. The device is used only for acquisition of EEG signals and may be used to log the events of interest.
  Other Names: NeuroSENSE Monitoring System, Model NS-701 (approved in Canada and European market (CE Mark)); NeuroFAST Monitoring System, Model NF-202 (US name, the device is not cleared by the FDA)
Other: Data collection — Non-invasive blood pressure (BP), heart rate (HR), respiratory rate (RR) and electroencephalogram (EEG) will be recorded during the surgery in all subjects. Also, information about all medically significant events, all study-related events (incl. patient's reactions, responses, observations and assessments) and administered medications (incl. end-tidal (ET) desflurane concentration) will be recorded along with time stamps.
  The anesthesia and physiological parameters (e.g., BP, HR, RR, ET agent concentration) outputted from the anesthesia monitor will be recorded electronically during the surgery by the anesthesia monitoring system (data-points will be recorded at least every 3 min for BP and every 10 sec for other variables).
  The EEG signal will be continuously recorded by NeuroSENSE NS-701 Monitor (described under a separate intervention).
  The CRC will also be present in the Operating Room (OR) to record and manage the recording of all the required information.
Other: Drug: Emergence by stepping down the desflurane ET — Anesthesia will be reduced to facilitate rapid recovery at the discretion of the anesthesiologist, about 20 minutes before the end of surgery. The desflurane ET will be stepped down from 0.8 MAC by steps of 0.2 MAC approximately every 5 min during the Emergence.
  Other Names: Suprane

SUMMARY:
The objective of this clinical study is to investigate whether the NeuroSENSE is an adequate monitor of hypnotic depth-of-anesthesia (DOA). Therefore, this study will investigate whether the information provided by the NeuroSENSE Monitor can help in assessing the hypnotic effect of anesthetics in adult patients undergoing general anesthesia.

DETAILED DESCRIPTION:
In particular, the study will focus on the correlation between the WAVcns index, a proprietary quantifier of cortical activity displayed by the NeuroSENSE, with (1) commonly assessed clinical endpoints/variables relating to the DOA, (2) changes in anesthetic drug administration, and (3) the anesthesiologist's assessment of the DOA based on standard of care monitors and his/her own observations of the patient state.

The hypothesis under evaluation is that the WAVcns index is an independent assessor of the progression of the anesthetic state and events of general anesthesia related to hypnotic endpoints.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years
* ASA (American Society of Anesthesiologist) physical status I, II, or III
* ability to read and understand the informed consent form
* undergoing anesthesia procedure requiring intubation
* scheduled to undergo either open or laparoscopic abdominal surgical procedures (e.g. colectomy, hysterectomy, radical retropubic prostatectomy, nephrectomy, pancreatectomy, etc.), breast surgery including reduction, reconstruction and mastectomies, or orthopedic surgeries under general anesthesia, expected to last at least 1 hour.

Exclusion Criteria:

* history of major head injury (possible abnormal EEG)
* acquired scalp or skull abnormalities (e.g. psoriasis, eczema, angioma, scar tissue, burr holes, cranial implants)
* evidence of recent trauma or active neurological disorder, stroke, seizure disorder, intellectual disability, dementia or diagnosis of Alzheimer's disease
* major antipsychotic medications taken within last 7 days (eg. Lithium, risperidone, olanzapine)
* known history of alcohol or drug abuse within last 30 days
* body mass index (weight in kilograms divided by square of height in meters) > 40.0 kg/m2
* uncontrolled hypertension with blood pressure recorded prior to surgery (systolic blood pressure > 200 mmHg or diastolic blood pressure > 110 mmHg)
* systolic blood pressure < 90 mmHg, recorded prior to surgery
* heart rate (HR) < 45 beats/min, recorded prior to surgery
* insulin-dependent diabetes mellitus
* pregnancy
* any serious medical condition that would interfere with cardiovascular response assessment or study results interpretation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing general anesthesia procedure in the context of either open or laparoscopic abdominal surgical procedures (e.g. colectomy, hysterectomy, radical retropubic prostatectomy, nephrectomy, pancreatectomy, etc.), breast surgery including reduction, reconstruction and mastectomies, or orthopedic surgeries under general anesthesia, expected to last at least 1 hour.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Prediction probability Pk for the WAVcns for consciousness vs unconsciousness | During induction of anesthesia, an expected average of 4 min
  The primary outcome will test the performance of WAVcns index in discriminating between consciousness and unconsciousness during induction of anesthesia. It will be evaluated using Receiver-Operating Characteristic (ROC), and Area Under Curve (AUC) will be calculated. Note that the AUC statistic is equal to the prediction probability Pk for dichotomous responses, such as consciousness and unconsciousness.

SECONDARY OUTCOMES:
Prediction probability Pk for the WAVcns for responders vs nonresponders to lidocaine aerosol | During induction of anesthesia, an expected average of 4 min
  This secondary outcome will test if the WAVcns index prior to lidocaine insufflations or intubation is a good predictor of patient response. The aerosolized lidocaine will be used as a standardized stimulus to objectively assess response observed at the larynx and seen in the patient during airway manipulation during induction of anesthesia.
Correlation of the WAVcns with primary anesthetic dosing | During anesthesia maintenance, an expected average of 2 hrs
  This secondary outcome will test if the WAVcns index during anesthesia maintenance correlates with primary anesthetic dosing (end tidal agent concentration).
Prediction probability for the WAVcns for responders vs nonresponders to verbal command | During emergence from anesthesia, an expected average of 20 min
  This secondary outcome will test if the WAVcns index accurately indicates return of consciousness (response to verbal command) during emergence.

OTHER OUTCOMES:
Correlation of the WAVcns with burst-suppression ratio | During maintenance of anesthesia, an expected average of 2 hrs
  This outcome will study the relationship between the WAVcns index and burst-suppression ratio during maintenance of anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Merchant, MD FRCPC, Principal Investigator — Fraser Health
Locations (2):
- Canada (2):
  - Fraser Health: Royal Columbian Hospital, New Westminster, British Columbia
  - Fraser Health: Eagle Ridge Hospital, Port Moody, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gorges M, West NC, Cooke EM, Pi S, Brant RF, Dumont GA, Ansermino JM, Merchant RN. Evaluating NeuroSENSE for assessing depth of hypnosis during desflurane anesthesia: an adaptive, randomized-controlled trial. Can J Anaesth. 2020 Mar;67(3):324-335. doi: 10.1007/s12630-019-01522-5. Epub 2019 Nov 5. PMID 31691253